CLINICAL TRIAL: NCT05969574
Title: Is Decreased Ovarian Reserve Related to an Increased Number of Previous Early Miscarriages? A Prospective Observational Study
Brief Title: Is Decreased Ovarian Reserve Related to an Increased Number of Previous Early Miscarriages?
Status: Recruiting | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Laura Melado, IVF Specialist, ART Fertility Clinics LLC
Other Study IDs: 2305-ABU-007-LM
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Infertility, Female; Miscarriage; Miscarriage, Recurrent; IVF
Keywords: miscarriage; infertility; IVF
MeSH Terms: conditions — Infertility, Female; Abortion, Spontaneous; Abortion, Habitual; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- AMH <1.3, at least 1 pregnancy or at least 1 miscarriage: Participants will not undergo any additional intervention compared to normal clinical assessment and routine testing of the ovarian reserve, which includes AMH and AFC. Investigators will follow standard stimulation protocols and medications.
  Interventions: Diagnostic Test: Transvaginal ultrasound; Diagnostic Test: Blood test AMH
- AMH <1.3, at least 1 pregnancy and no miscarriage: Participants will not undergo any additional intervention compared to normal clinical assessment and routine testing of the ovarian reserve, which includes AMH and AFC. Investigators will follow standard stimulation protocols and medications.
  Interventions: Diagnostic Test: Transvaginal ultrasound; Diagnostic Test: Blood test AMH
- AMH ≥ 1.3, at least 1 pregnancy or at least 1 miscarriage: Participants will not undergo any additional intervention compared to normal clinical assessment and routine testing of the ovarian reserve, which includes AMH and AFC. Investigators will follow standard stimulation protocols and medications.ons.
  Interventions: Diagnostic Test: Transvaginal ultrasound; Diagnostic Test: Blood test AMH
- AMH ≥1.3, at least 1 pregnancy and no miscarriage: Participants will not undergo any additional intervention compared to normal clinical assessment and routine testing of the ovarian reserve, which includes AMH and AFC. Investigators will follow standard stimulation protocols and medications.
  Interventions: Diagnostic Test: Transvaginal ultrasound; Diagnostic Test: Blood test AMH

INTERVENTIONS:
Diagnostic Test: Transvaginal ultrasound — Transvaginal ultrasound for antral follicle count (AFC) performed on the day of first consultation
Diagnostic Test: Blood test AMH — Measurement of AMH performed on the day of first consultation

SUMMARY:
This study aims to explore the potential correlation between decreased ovarian reserve and previous history of early miscarriage.

DETAILED DESCRIPTION:
By investigating the prevalence of low ovarian reserve (LOR) in populations with specific reproductive histories (such as recurrent pregnancy loss, G0, and ectopic pregnancy), as well as the aneuploidy rates of embryos produced with Preimplantation Genetic Testing for Aneuploidies (PGT-A), Investigators can better understand how LOR impacts fertility outcomes in these populations. This information can be used to inform clinical decision-making, such as whether participants with LOR should consider alternative or whether they would benefit from additional interventions to improve ovarian function.

Ultimately, by improving our understanding of how LOR impacts fertility outcomes in specific populations, Investigators can help to improve the overall success rates of infertility treatment, reduce anxiety, and distress, and help participants achieve goals of becoming parents.

ELIGIBILITY:
Inclusion Criteria:

1. All participants with at least 1 previous pregnancy, who are assessed in one of our clinics (ART Fertility Clinics Abu Dhabi, Al Ain, Dubai)

Exclusion Criteria:

1. Severe male factor (azoospermia, cryptozoospermia, severe oligoasthenoteratozoospermia (OAT))
2. Severe Endometriosis and adenomyosis based on positive anamnesis or ultrasound performed in our center during the first consultation
3. Uterine abnormalities (e.g. fibroids, different degrees of uterine septum), diagnosed by ultrasound
4. History of ovarian surgery, chemotherapy, or radiation therapy
5. Known genetic disorder or chromosomal abnormality
6. BMI >40Kg/m2
7. Currently using hormonal contraception or hormone replacement therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: All participants who visit ART Fertility clinics in Abu Dhabi, Al Ain and Dubai for first consultation
Sampling Method: Non-Probability Sample
Enrollment: 2059 (Estimated)
Dates: Start 2023-09-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
AMH | 1 day
  Anti-Müllerian Hormone Test
AFC | 1 day
  Antral follicle count

CONTACTS AND LOCATIONS:
Overall Officials: Laura Melado, PhD, Principal Investigator — ART Fertility Clinics LLC
Locations (3):
- United Arab Emirates (3):
  - ART Fertility Clinics LLC, Abu Dhabi, Abu Dhabi Emirate
  - ART Fertility Clinics Al Ain, Al Ain City
  - ART Fertility Clinics Dubai, Dubai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ESHRE working group on Ectopic Pregnancy; Kirk E, Ankum P, Jakab A, Le Clef N, Ludwin A, Small R, Tellum T, Toyli M, Van den Bosch T, Jurkovic D. Terminology for describing normally sited and ectopic pregnancies on ultrasound: ESHRE recommendations for good practice. Hum Reprod Open. 2020 Dec 16;2020(4):hoaa055. doi: 10.1093/hropen/hoaa055. eCollection 2020. PMID 33354626
- [Background] Tan J, Luo L, Jiang J, Yan N, Wang Q. Decreased Ovarian Reserves With an Increasing Number of Previous Early Miscarriages: A Retrospective Analysis. Front Endocrinol (Lausanne). 2022 Jun 10;13:859332. doi: 10.3389/fendo.2022.859332. eCollection 2022. PMID 35757430
- [Background] Bliddal S, Feldt-Rasmussen U, Forman JL, Hilsted LM, Larsen EC, Christiansen OB, Nielsen CH, Kolte AM, Nielsen HS. Anti-Mullerian hormone and live birth in unexplained recurrent pregnancy loss. Reprod Biomed Online. 2023 Jun;46(6):995-1003. doi: 10.1016/j.rbmo.2023.01.023. Epub 2023 Feb 3. PMID 37055255
- [Background] Stirrat GM. Recurrent miscarriage. II: Clinical associations, causes, and management. Lancet. 1990 Sep 22;336(8717):728-33. doi: 10.1016/0140-6736(90)92215-4. PMID 1975901
- [Background] Wang X, Chen C, Wang L, Chen D, Guang W, French J. Conception, early pregnancy loss, and time to clinical pregnancy: a population-based prospective study. Fertil Steril. 2003 Mar;79(3):577-84. doi: 10.1016/s0015-0282(02)04694-0. PMID 12620443
- [Background] Coomarasamy A, Dhillon-Smith RK, Papadopoulou A, Al-Memar M, Brewin J, Abrahams VM, Maheshwari A, Christiansen OB, Stephenson MD, Goddijn M, Oladapo OT, Wijeyaratne CN, Bick D, Shehata H, Small R, Bennett PR, Regan L, Rai R, Bourne T, Kaur R, Pickering O, Brosens JJ, Devall AJ, Gallos ID, Quenby S. Recurrent miscarriage: evidence to accelerate action. Lancet. 2021 May 1;397(10285):1675-1682. doi: 10.1016/S0140-6736(21)00681-4. Epub 2021 Apr 27. PMID 33915096
- [Background] Bunnewell SJ, Honess ER, Karia AM, Keay SD, Al Wattar BH, Quenby S. Diminished ovarian reserve in recurrent pregnancy loss: a systematic review and meta-analysis. Fertil Steril. 2020 Apr;113(4):818-827.e3. doi: 10.1016/j.fertnstert.2019.11.014. Epub 2020 Mar 4. PMID 32145928
- [Background] Seifer DB. Connecting the dots between oocyte quantity and quality in diminished ovarian reserve. Fertil Steril. 2021 Apr;115(4):890. doi: 10.1016/j.fertnstert.2021.01.020. Epub 2021 Mar 6. No abstract available. PMID 33750616
- [Background] Tarasconi B, Tadros T, Ayoubi JM, Belloc S, de Ziegler D, Fanchin R. Serum antimullerian hormone levels are independently related to miscarriage rates after in vitro fertilization-embryo transfer. Fertil Steril. 2017 Sep;108(3):518-524. doi: 10.1016/j.fertnstert.2017.07.001. PMID 28865551
- [Background] Lyttle Schumacher BM, Jukic AMZ, Steiner AZ. Antimullerian hormone as a risk factor for miscarriage in naturally conceived pregnancies. Fertil Steril. 2018 Jun;109(6):1065-1071.e1. doi: 10.1016/j.fertnstert.2018.01.039. Epub 2018 Jun 2. PMID 29871793
- [Background] Atasever M, Soyman Z, Demirel E, Gencdal S, Kelekci S. Diminished ovarian reserve: is it a neglected cause in the assessment of recurrent miscarriage? A cohort study. Fertil Steril. 2016 May;105(5):1236-1240. doi: 10.1016/j.fertnstert.2016.01.001. Epub 2016 Jan 21. PMID 26806685
- [Background] Leclercq E, de Saint Martin L, Bohec C, Le Martelot MT, Roche S, Alavi Z, Mottier D, Pasquier E. Blood anti-Mullerian hormone is a possible determinant of recurrent early miscarriage, yet not conclusive in predicting a further miscarriage. Reprod Biomed Online. 2019 Aug;39(2):304-311. doi: 10.1016/j.rbmo.2019.04.004. Epub 2019 Apr 12. PMID 31186176
- [Background] Jaswa EG, McCulloch CE, Simbulan R, Cedars MI, Rosen MP. Diminished ovarian reserve is associated with reduced euploid rates via preimplantation genetic testing for aneuploidy independently from age: evidence for concomitant reduction in oocyte quality with quantity. Fertil Steril. 2021 Apr;115(4):966-973. doi: 10.1016/j.fertnstert.2020.10.051. Epub 2021 Feb 12. PMID 33583594